CLINICAL TRIAL: NCT05266196
Title: A Rollover Protocol to Allow for Continued Access to the LSD1 Inhibitor Seclidemstat (SP-2577)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Salarius Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALA-004-RO21
Record Dates: First submitted 2021-11-11; First posted 2022-03-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Ewing Sarcoma; Myxoid Liposarcoma; Desmoplastic Small Round Cell Tumor; Extraskeletal Myxoid Chondrosarcoma; Angiomatoid Fibrous Histiocytoma; Clear Cell Sarcoma; Myoepithelial Tumor; Low Grade Fibromyxoid Sarcoma; Sclerosing Epithelioid Fibrosarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Liposarcoma, Myxoid; Desmoplastic Small Round Cell Tumor; Chondrosarcoma, Extraskeletal Myxoid; Histiocytoma, Angiomatoid Fibrous; Sarcoma, Clear Cell; Myoepithelioma | interventions — seclidemstat; Topotecan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single agent (Experimental): Single agent seclidemstat, as assigned per parent protocol
  Interventions: Drug: Seclidemstat
- TC Combination (Experimental): Combination of seclidemstat with topotecan and cyclophosphamide, as assigned per parent protocol
  Interventions: Drug: Seclidemstat

INTERVENTIONS:
Drug: Seclidemstat — Treatment assigned as per parent protocol
  Other Names: topotecan; cyclophosphamide

SUMMARY:
This rollover protocol allows continued access to seclidemstat (SP-2577) for patients who are still receiving clinical benefit on completed or closed Salarius sponsored studies.

DETAILED DESCRIPTION:
The population for the rollover study should be consistent with the population defined in the parent study. The primary eligibility criteria for a patient to enter the rollover protocol is the participation and completion of a Salarius sponsored study with seclidemstat. Safety data and an evaluation of anti-tumor activity will be collected.

Patients who have completed a prior study with seclidemstat and who are assessed by the Investigator to continue to benefit from ongoing treatment will be eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently enrolled in a Salarius-sponsored study that is approved to enroll into this rollover study, and are receiving seclidemstat as monotherapy or in combination with other study treatment per the parent protocol (i.e. topotecan and cyclophosphamide). The maximum time between discontinuing the parent protocol and starting this rollover protocol is 14 days.
2. Patient is currently benefiting from the treatment with seclidemstat monotherapy or combination treatment, as determined by the investigator
3. Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements
4. Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures
5. Ability to understand and the willingness to sign a written informed consent document.
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of seclidemstat administration.

Exclusion Criteria:

1. Patient has been permanently discontinued from study treatment in the parent study due to any reason, except for the purpose of entering this open label rollover study.
2. Pregnant and breastfeeding women are excluded from this study. The effects of seclidemstat on the developing human fetus have the potential for teratogenic or abortifacient effects. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with seclidemstat.
3. Patient is receiving prohibited concomitant therapy as described in Section 5.4.2 of the rollover protocol, or therapy not allowed in the parent protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Length of time receiving study treatment | months on study where patients continue to receive clinical benefit, up to 5 years
  Length of time receiving treatment with seclidemstat as single agent or in combination with assigned parent protocol therapy

SECONDARY OUTCOMES:
Number of patients enrolled through study completion | Number of patients enrolled on study who continue to receive clinical benefit, up to 5 years
  Number of patients enrolled who received seclidemstat
Evaluate safety & tolerability utilizing the most current version of CTCAE | During treatment while on study and continuing to receive clinical benefit, up to 5 years
  Evaluate the safety and tolerability of seclidemstat by characterizing adverse events according to the most current version of CTCAE
Evaluate anti-tumor activity based upon imaging studies according to RECIST v1.1 | During treatment while on study and continuing to receive clinical benefit, up to 5 years
  Evaluate the anti-tumor activity of seclidemstat based upon imaging studies according to RECIST v1.1

OTHER OUTCOMES:
Assess PK profile, maximum plasma concentration (Cmax) | During treatment while on study and continuing to receive clinical benefit, up to 5 years
  • To assess pharmacokinetics of seclidemstat and metabolites in post-treatment tumor biopsies to compare partitioning of these analytes between tumor and plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No